CLINICAL TRIAL: NCT00871234
Title: Effects of Etravirine (INTELENCETM) on Endothelial Function in HIV-uninfected Adults: A Pilot Study
Brief Title: Effects of Etravirine on Endothelial Function in HIV-uninfected Adults: A Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Tibotec Therapeutics, a Division of Ortho Biotech Products, L.P., USA (Industry)
Responsible Party: Samir K. Gupta, MD, MS, Indiana University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 0812-18 (TMC125HIV4003)
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Results first posted 2011-01-05 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2010-12

CONDITIONS: Endothelial Function; Lipids; Insulin Resistance; Inflammation; HIV Infections
Keywords: HIV; Endothelial function; Etravirine
MeSH Terms: conditions — Insulin Resistance; Inflammation; HIV Infections | interventions — etravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Etravirine — Two one-hundred mg tablets orally twice daily for four weeks
  Other Names: INTELENCETM

SUMMARY:
The purpose of this study is to determine the safety and effects of etravirine, an HIV antiretroviral medication, on vascular function.

DETAILED DESCRIPTION:
We hypothesize that in HIV-uninfected subjects, etravirine 200mg twice daily for four weeks will have no effect on endothelial function. The primary objective of this study is to determine the effects of etravirine 200mg twice daily given for four weeks on endothelial function, measured as flow-mediated dilation (FMD) of the brachial artery, in HIV-uninfected subjects. Secondary objectives include determination of the effects of etravirine 200mg twice daily given for four weeks on safety measures, lipid fractions, HOMA-IR, blood pressure, inflammatory parameters, and endothelial activation parameters.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Negative ELISA for HIV-1 or HIV-2 at screening
3. Negative hepatitis B surface antigen at screening
4. Negative hepatitis C antibody at screening
5. For women of reproductive potential, a negative urine pregnancy test at screening and willingness to use two forms of birth control during the course of the study
6. No history of diabetes, hypertension, or dyslipidemia
7. No anticipated changes or additions to other medical therapies during the course of the study

Exclusion Criteria:

1. Inability to provide written, informed consent
2. Known allergy/intolerance to etravirine or nitroglycerin
3. Absolute neutrophil count < 750cell/mL at screening
4. Hemoglobin <11g/dL at screening
5. Platelet count <100,000/mL at screening
6. Estimated creatinine clearance (per Cockcroft-Gault equation) <55 mL/min at screening
7. Liver transaminases (AST or ALT) > 100 IU/mL or total bilirubin > 1.5mg/dL at screening
8. Breastfeeding at screening and during the course of the study
9. Hypotension, defined as SBP<90mmHg at time of each main study visit before brachial artery ultrasound measurements
10. Receipt of investigational agents, cytotoxic chemotherapy, systemic glucocorticoids (>10mg/day of prednisone or the equivalent), or anabolic steroids within 30 days of each screening visit or each main study visit
11. Use of sildenafil (Viagra or Silagra), vardenafil (Levitra), or tadalafil (Cialis), within 72 hours (before or after) of brachial artery reactivity testing
12. Indwelling vascular catheters within any upper body vessel at time of brachial artery reactivity testing
13. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements
14. Acute therapy for serious infection or other serious medical illnesses (in the judgment of the site investigator) requiring systemic treatment and/or hospitalization within 14 days prior to each screening and study visit
15. History of migraine headaches
16. History of Raynaud's phenomenon
17. History of cardiac arrythmias
18. History of hypothyroidism or hyperthyroidism that is untreated (defined as a TSH outside the normal range on most recent testing during normal clinical care)
19. History of carotid bruits.
20. History of any tobacco use (cigarette smoking, cigar smoking, chewing tobacco) or nicotine replacement treatments (patch, gum) within one year of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-04; Primary Completion 2010-03 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir K Gupta, MD, MS, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Infectious Diseases Research Center, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between April 2009 and March 2010. Participants were recruited via advertisements and word-of-mouth.
Pre-assignment Details: After participant enrollment, a screening visit was performed to determine eligibility. Participants may have been excluded from entering the study if they were found to be ineligible.
Groups:
- Etravirine: Healthy volunteers receiving etravirine 200mg orally twice daily
Period: Overall Study
Arm/Group | Etravirine
Started | 28
Completed | 23
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Etravirine
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Age Continuous [Median (Inter-Quartile Range); unit: years] | 40 [28 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Flow-mediated Dilation (FMD) of the Brachial Artery
Description: FMD is measured as the percentage increase in brachial artery diameter after increase in blood flow. We measured the change in this percentage from entry (before etravirine was started) and again at four weeks after receiving etravirine.
Time Frame: Entry and four weeks
Population: FMD analysis was per protocol restricted to those who completed the four week trial. The safety analysis was ITT.
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Etravirine
Number analyzed (Participants) | 28
Percentage | 0.03 [-3.21 to 0.97]
Statistical Analysis 1: Comparison: Etravirine; Test type: Superiority or Other; p = 0.36, Wilcoxon signed-rank; Median Difference (Net) = 0.03

2. Secondary Outcome: Lipid Fractions
Time Frame: Four weeks
Reporting Status: Not Posted

3. Secondary Outcome: Insulin Sensitivity [(Homeostasis Model Assessment-Insulin Resistance (HOMA-IR)]
Time Frame: Four weeks
Reporting Status: Not Posted

4. Secondary Outcome: Blood Pressure
Time Frame: Four weeks
Reporting Status: Not Posted

5. Secondary Outcome: Inflammatory Biomarkers
Time Frame: Four weeks
Reporting Status: Not Posted

6. Secondary Outcome: Endothelial Activation Biomarkers
Time Frame: Four weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Six weeks
Arm/Group | Etravirine
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 15/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Etravirine (N=28)
Neuropathic tingling or pain (Nervous system disorders) | 2 (2) — Both Grade 1; both resolved spontaneously within 3 days and were not treatment limiting.
Rash (Skin and subcutaneous tissue disorders) | 2 (2) — Both Grade 2; both resolved within 3 days upon discontinuation of study drug.
Diarrhea (Gastrointestinal disorders) | 2 (2) — Both Grade 1; both resolved spontaneously within 11 days and were not treatment limiting.
Nausea/vomiting (Gastrointestinal disorders) | 2 (2) — Both Grade 1; both resolved spontaneously within 2 days and were not treatment limiting.
Constipation (Gastrointestinal disorders) | 3 (3) — All Grade 1; all resolved spontaneously within 11 days and were not treatment limiting.
Headache (Nervous system disorders) | 4 (4) — All Grade 1; all spontaneously resolved within 12 days and were not treatment-limiting.
Dizziness (Nervous system disorders) | 2 (2) — Both Grade 1; both resolved spontaneously within 2 days and were not treatment limiting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No